CLINICAL TRIAL: NCT05849025
Title: Invasive Hemodynamic Control Cohort for The Mayo Clinic Adult Congenital Heart Disease (MACHD) Registry
Brief Title: A Study of Invasive Hemodynamic for MACHD Registry
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Other Study IDs: 23-001939; R01HL160761 (NIH)
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study is being done to provide comparative data to the Mayo Clinic Adult Congenital Heart Disease Registry.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to Consent
* BMI </= 30
* Systolic BP </= 140mmHg
* Diastolic BP </= 90
* eGFR > 30 (within prior 3 months) to confirm kidney function
* Able to undergo an MRI

Exclusion Criteria:

* History of Cardiovascular disease that may affect the results of the testing performed.
* Any Current orthopedic limitations
* Currently taking any cardiac medication
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals without cardiac conditions will be recruited from Mayo Clinic in Rochester, MN.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular reserve | Baseline
  The slope of mean pulmonary artery pressure / cardiac output (mPAP/CO)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No